CLINICAL TRIAL: NCT02542969
Title: A Single Center, Open-label, Drug Interaction Study of MGL-3196 With Rosuvastatin and Simvastatin in Healthy Subjects
Brief Title: Drug Interaction Study of MGL-3196 With Rosuvastatin and Simvastatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Madrigal Pharmaceuticals, Inc. (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MGL-3196-03
Record Dates: First submitted 2015-09-04; First posted 2015-09-07 (Estimated); Last update posted 2022-09-02 (Actual); Status verified 2015-09

CONDITIONS: Healthy
MeSH Terms: interventions — Simvastatin; Rosuvastatin Calcium; resmetirom

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Other): Simvastatin followed by Rosuvastatin then MGL-3196 daily followed by separate co-administration of Simvastatin and Rosuvastatin
  Interventions: Drug: Simvastatin; Drug: Rosuvastatin; Drug: MGL-3196

INTERVENTIONS:
Drug: Simvastatin
  Other Names: Zocor
Drug: Rosuvastatin
  Other Names: Crestor
Drug: MGL-3196
  Other Names: VIA-3196

SUMMARY:
The purpose of this study is to determine whether MGL-3196 alters the pharmacokinetics of rosuvastatin and/or simvastatin in healthy male subjects and female subjects not of child-bearing potential.

ELIGIBILITY:
Inclusion Criteria:

* Must be willing and able to provide written informed consent.
* Healthy, non-smoking, male or female between the ages of 18 and 55 years (inclusive).
* Body weight > 50 kg and BMI between 18 and 32 kg/m2 (inclusive).
* If female, is of non-child bearing potential (i.e., surgically [bilateral oophorectomy, hysterectomy, hysteroscopic sterilization, or tubal ligation]. Or, is naturally sterile [>12 consecutive months without menses]) with verification by follicle stimulating hormone (FSH) at screening.
* If male and non-vasectomized, must agree to use a condom with spermicide or abstain from sexual intercourse during the study until 30 days beyond the last dose of study drug. No restrictions are required for a vasectomized male provided his vasectomy has been performed 4 months or more prior to first dose of study drug. A male who has been vasectomized less than 4 months prior to study start must follow the same procedure as a non-vasectomized male.

Exclusion Criteria:

* Any clinically significant abnormal findings during physical examination including blood pressure, heart rate or rhythm, clinical laboratory tests or 12-lead ECG.
* Evidence or history of clinically significant hematological, endocrine, pulmonary, gastrointestinal, cardiovascular, renal, hepatic, neurological or psychiatric disease.
* Thyroid stimulating hormone test at screening outside the normal range. Repeat testing is allowed once at the discretion of the Investigator.
* Current or recent (<6 months) hepatobiliary disease; or aspartate aminotransferase (AST), alanine aminotransferase (ALT) or direct bilirubin greater than the upper limit of reference range at screening. Repeat testing is allowed once at the discretion of the Investigator.
* Elevated creatine kinase (CK) at screening (one repeat test allowed).
* Gilbert's syndrome.
* Positive screening test for HIV antibody, Hepatitis B surface antigen or Hepatitis C antibody.
* Abnormal screening ECG: including machine-read QTc >450 msec (confirmed by manual over read), QRS >110 msec, intermittent bundle branch block, frequent premature atrial or premature ventricular contractions, or any rhythm other than normal sinus rhythm which is interpreted by the Investigator to be clinically significant.
* History of sensitivity to a similar study drug (e.g., Karo Bio KB2115 or Metabasis MB7811), or a history of important drug or other allergy (except for untreated, asymptomatic seasonal allergies at time of dosing) unless deemed not clinically significant by the Investigator.
* History of sensitivity to thyroid medication.
* History of intolerance to or adverse reaction to a statin, or history of myopathy including rhabdomyolysis.
* Intolerance to beta-blockers (beta-blocker treatment could be appropriate to alleviate tachycardia if observed).
* Participation in another clinical trial of an investigational drug (or medical device) within the last 30 days prior to the first dosing day, or who have been exposed to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of St. John's Wort within 28 days before the first dose of study drug.
* Unwilling to forgo consumption of red wine, Seville oranges, grapefruit or grapefruit juice and/or pomelos, star fruit, grapefruit hybrids or other citrus juices from 5 days prior to the first dose of study drug and throughout the study.
* Subjects with a history of drug or alcohol abuse as defined by the Diagnostic and Statistical Manual 5th Edition.
* History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for men (1 drink = 5 ounces of wine or 12 ounces of beer or 1.5 ounces of hard liquor) within 6 months prior to screening.
* Use of acetaminophen within 7 days before dosing and throughout the study except for the treatment of an adverse event as directed by the Investigator.
* History of regular use of tobacco or nicotine containing products within the past 6 months relative to screening.
* Positive urine drug screen or alcohol test at screening or Day -1.
* Women who are pregnant or may become pregnant, or are nursing.
* Strenuous physical activity which could cause muscle aches or injury, including contact sports, at any time from 3 days prior to first dose of study drug until completion of the study.
* Excessive caffeine intake (>3 cups of coffee/day or equivalent).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2015-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Area under the curve from the time of dosing extrapolated to infinity (AUC(0-inf)) of Rosuvastatin as affected by MGL-3196 | 72 hours
AUC(0-inf) of Simvastatin as affected by MGL-3196 | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Gerri Poss, MD, Principal Investigator — Celerion
Locations (1):
- Celerion, Tempe, Arizona, United States